CLINICAL TRIAL: NCT04825457
Title: Comparative Study of Anchoring-tip vs. Conventional EMR of Intermediate-Size Colorectal Polyps: Multi-center, Prospective, Randomized Controlled Trial
Brief Title: Comparative Study of Anchoring-tip vs. Conventional EMR of Colorectal Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Chilgok Hospital (Other)
Responsible Party: Principal Investigator, Joon Seop Lee, Clinical Assistant Professor, Kyungpook National University Chilgok Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-10-008
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Polyp

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anchoring-tip EMR (Active Comparator): AEMR, the snare tip was projected from the sheath by 1-2 mm length. Consequently, a small mucosal incision was made at proximal side of lesion. Then the snare was deployed progressively and adjusted around the lesion trying to obtain free margins.
  Interventions: Procedure: Anchoring-tip vs. Conventional
- Conventional EMR (Active Comparator): After injection of normal saline solution mix, snaring was tried for CEMR.
  Interventions: Procedure: Anchoring-tip vs. Conventional

INTERVENTIONS:
Procedure: Anchoring-tip vs. Conventional — Anchoring-tip: the snare tip was projected from the sheath by 1-2 mm length. Consequently, a small mucosal incision was made at proximal side of lesion. Then the snare was deployed progressively and adjusted around the lesion trying to obtain free margins. At the final step of both conventional and Tip-in EMR, the lesion was resected.
  Conventional: After injection of normal saline solution mix, snaring was tried for polyp resection.

SUMMARY:
Endoscopic mucosal resection (EMR) is an effective and has been widely used technique for the treatment of superficial colorectal neoplasms. Although, conventional EMR (CEMR) showed high efficacy for the management of colorectal superficial neoplasms, there is problematic limitation in this technique - incomplete resection. In literature, the anchoring-tip EMR (AEMR), named as "Tip-in EMR" was first introduced in 2016 from Japan. Recently, several retrospective studies have been suggested about the effectiveness of AEMR. However, there has been no prospective randomized controlled study to identify its advantage over CEMR. Therefore, the investigators performed a multicenter randomized controlled trial to estimate the effectiveness of AEMR compared with CEMR for the endoscopic treatment of intermediate-size (10 to 20 mm) colorectal polyps.

DETAILED DESCRIPTION:
After injection of normal saline solution mix, snaring was tried for CEMR. In AEMR, the snare tip was projected from the sheath by 1-2 mm length. Consequently, a small mucosal incision was made at proximal side of lesion. Then the snare was deployed progressively and adjusted around the lesion trying to obtain free margins. At the final step of both conventional and Tip-in EMR, the lesion was resected.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate-size (10 to 20 mm) colorectal polyps
* Morphologically sessile (Is), slightly elevated (IIa), flat (IIb), and slightly depressed (IIc) as Paris classification of superficial neoplastic lesions
* Laterally spreading tumor (granular and nongranular type) as Kudo classification.

Exclusion Criteria:

* Pedunculated or excavated/ulcerated polyps
* Polyps with features strongly suggestive of submucosal invasive carcinoma
* Polyps in patients with inflammatory bowel disease, familial polyposis, electrolyte abnormality, and coagulopathy
* Residual lesions after endoscopic resection or presence of severe submucosal fibrosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Primary outcome was comparing the R0 resection rate between Anchoring-tip EMR and Conventional EMR. | From EMR to reporting of histopathology, 1 month
  Histopathologic complete resection (R0) was defined as en bloc resection and clear lateral and vertical resection margins.

CONTACTS AND LOCATIONS:
Locations (1):
- Joon Seop Lee, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No